CLINICAL TRIAL: NCT00007826
Title: A Phase I/II Trial of an Allogeneic Cell Based Vaccine and an Anti-Idiotypic Antibody Vaccine Approach for Metastatic Adenocarcinoma of the Colon or Rectum
Brief Title: Monoclonal Antibody Therapy and/or Vaccine Therapy in Treating Patients With Locally Advanced or Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Onyvax (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068071; ONYVAX-SGCRO01; NCI-V00-1599
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2005-02

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — BCG Vaccine; Aluminum Hydroxide

INTERVENTIONS:
Biological: BCG vaccine
Biological: monoclonal antibody 105AD7 anti-idiotype vaccine
Drug: alum adjuvant

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Vaccines made from cancer cells may make the body build an immune response to kill colorectal tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of monoclonal antibody therapy and/or vaccine therapy in treating patients who have locally advanced or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of monoclonal antibody 105AD7 anti-idiotypic vaccine and ONYCR1, ONYCR2, and ONYCR3 allogeneic adenocarcinoma cell-based vaccines in patients with locally advanced or metastatic adenocarcinoma of the colon or rectum.
* Determine any immunological response to these treatment regimens in these patients.
* Determine the 6-month and 1-year survival of these patients after receiving these treatment regimens.
* Determine the tumor response to these treatment regimens in these patients.

OUTLINE: This is an open-label study. Patients are assigned to one of three treatment arms.

* Arm I: Patients receive monoclonal antibody 105AD7 anti-idiotype vaccine (MOAB 105AD7) plus BCG intradermally (ID) weekly for weeks 1 and 2; MOAB 105AD7 ID plus alum adjuvant intramuscularly (IM) weekly for weeks 4 and 6; and then MOAB 105AD7 ID alone monthly for up to 12 months.
* Arm II: Patients receive ONYCR1, ONYCR2, and ONYCR3 allogeneic adenocarcinoma cell-based vaccines plus BCG ID weekly for weeks 1 and 2; these vaccines ID weekly for weeks 4 and 6, and then monthly for up to 12 months.
* Arm III: Patients receive MOAB 105AD7, ONYCR1, ONYCR2, and ONYCR3 allogeneic adenocarcinoma cell-based vaccines, and BCG ID weekly for weeks 1 and 2; MOAB 105AD7 and ONYCR1, ONYCR2, and ONYCR3 allogeneic adenocarcinoma cell-based vaccines ID plus alum adjuvant IM weekly for weeks 4 and 6; and then MOAB 105AD7 and ONYCR1, ONYCR2, and ONYCR3 allogeneic adenocarcinoma cell-based vaccines monthly for up to 12 months.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 45 patients (15 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed locally advanced or metastatic adenocarcinoma of the colon or rectum

  * Not amenable to curative surgery and either refractory to or inappropriate for chemotherapy
  * Patient must have received adequate or appropriate prior chemotherapy for metastatic disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other prior malignancy within the past 5 years except adequately treated basal cell carcinoma of the skin or carcinoma in situ
* No history of immunodeficiency
* No concurrent unstable medical condition that would preclude study
* No psychological, familial, sociological, or geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 month since prior immunomodulatory drugs

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* At least 1 month since prior corticosteroids
* No concurrent corticosteroids

Radiotherapy:

* At least 6 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics

Other:

* At least 4 weeks since other prior anticancer drug
* No other concurrent investigational anticancer agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-04

CONTACTS AND LOCATIONS:
Overall Officials: Fiona J. Lofts, MD, Study Chair — St. George's Hospital
Locations (1):
- St. George's Hospital, London, England, United Kingdom